CLINICAL TRIAL: NCT01340222
Title: Evaluation of the Prognostic Value of Monocytes and Lymphocyte Phenotyping, Along With Intracellular MCP-1 Expression, to Predict Preterm Delivery for Women Hospitalized for Threat of Preterm Labor Between 24 and 34 Weeks of Amenorrhea: PhenoMAP Study
Brief Title: Monocyte Chemotactic Protein-1 (MCP-1) Expressing Monocytes to Predict Preterm Delivery: PhenoMAP Study
Acronym: PHENOMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SAGOT PHRC IR 2010
Record Dates: First submitted 2011-04-19; First posted 2011-04-22 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Preterm Labour
Keywords: Preterm labour; monocyte; lymphocyte; MCP-1; Treg Lymphocytes; biologic markers; immunology; HLA-DR; Th17
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients (Other)
  Interventions: Biological: biological samples
- Volunteers (Other)
  Interventions: Biological: biological samples

INTERVENTIONS:
Biological: biological samples — 4 blood sampling will be made at J0, J2, J4, J6 befor delivery and 1 blood sampling 3 days after delivery

SUMMARY:
The threat of preterm labour (PTL) is the first cause of hospitalization in the course of pregnancy. Its diagnostic is based on clinical examination with a positive predictive value of about 40 %. The role of the Monocyte chemotactic protein-1 (MCP-1) in delivery has been suggested by its secretion in the amniotic fluid during labour and by the increase in the expression of its RNA messengers in the peripheral maternal blood. We have also shown that the proportion of MCP-1-expressing monocytes is higher in women with vaginal delivery compared with those with caesarean delivery prior the onset of labour.

OBJECTIVES : Primary To seek link between the respective proportions of circulating maternal monocyte and lymphocyte subpopulations and the true onset of PTL characterised by delivery occurring within 7 days post admission. Secondary: to (1) compare the predictive values of these new markers with those currently used, e.g. quantification of fœtal fibronectin and assessment of cervical length and effacement, (2) Compare the respective proportions of monocytes and lymphocyte subpopulations in maternal blood and fœtal membranes, (3) determine if a correlation exists between the activation markers expressed by maternal monocyte and lymphocyte subpopulations and the neonatal outcomes of preterm infants.

MATERIAL AND METHODS: 200 patients with a singleton pregnancy between 24 and 34 weeks of amenorrhea and complicated PTL, will be prospectively included in the maternity wards of Galway (Ireland) and of Dijon with the support of the perinatal network of Burgundy. A 2X5ml blood sample will be collected upon admission, at D1, D2, D4 and D6 for women who did not deliver within the first 7 days; finally, another blood sample will be drawn upon discharge. After delivery, foetal membranes will be collected to characterize and compare the various monocyte and lymphocyte subpopulations in the maternal blood. The characterization and the study of the level of activation of blood and foetal membrane cells will be performed using flow cytometry technique with suitable markers. The main judgment criteria will be the percentage of monocytes positively expressing MCP-1 for all three monocyte subpopulations ("inflammatory", "residents or patrollers" and "intermediates", according to CD14, CD16, CCR2 and MCP-1 markers. Lymphocyte subpopulations will be assessed using the following markers: CD45, CD3, CD4, CD8 (T lymphocytes), HLA-DR (activated T lymphocytes), CD19 (B lymphocytes), CD16/CD56 (NK Cells), intracellular IFN-gamma (Th1 lymphocytes), intracellular IL-4 (Th-2 lymphocytes), intracellular IL-17 and CCR6 (Th17 lymphocytes), CD4, CD25, Foxp3 and CD127 (Tregs). Univariate statistical analysis of quantitative data will be performed using the Mann and Witney test or ANOVA, after verification of the conditions of application. The comparisons of percentages will be done using Chi-square Pearson tests and the Fisher's exact test, as appropriate. The multivariate analysis will be performed using a stepwise descending analysis.

TRANSLATIONAL DIMENSION: The characterization of the various monocyte and lymphocyte subpopulations in the maternal blood and in the foetal membranes might constitute an " immunological signature " of the labour and therefore validate the relevance of a predictive marker for clinicians.

EXPECTED RESULTS AND PERSPECTIVES: The study of the various monocyte and lymphocyte subpopulations in the maternal blood will allow to better characterise the immunological mechanisms occurring at the start of premature labour and to identity predictive markers of the preterm delivery, to validate prospectively in order to optimize the management of PTL

ELIGIBILITY:
Inclusion Criteria for patients:

* Threat of preterm labour (PTL) occurring between 24 and 34 WOA, defined according to validated criteria i.e. by (1) the presence of regular uterine contractions, lasting at least 30 seconds at a frequency ≥ 4 contractions every 30 minutes and confirmed by an external tocogram, (2) a cervical dilation of 3 cm or greater, to focus on true preterm labour, for the nulliparous women and 1-3 cm among primiparous women or multiparous and (3) a cervical obliteration >50%, or a cervix less than 25mm according to the echography, when this information is available. The first two criteria being mandatory, the third one optional as it is more subjective, or less likely to be available for every patient.

  * Person who has given written consent
  * Singleton pregnancy

Inclusion Criteria for volunteers:

* Person who has given written consent
* Group 1: Women of reproductive age who have never had a pregnancy, even if not completed to term.
* Group 2: Single full-term, uncomplicated pregnancy (= out of hospital) older than 6 months.

Exclusion Criteria for patients:

* Pre-existing diabetes or gestational diabetes, morbid obesity (BMI > 35 kg/m2) as these situations modify the expression of MCP-1.
* Woman presenting a spontaneous rupture of membranes (SRM) with confirmed or probable chorioamniotitis
* Inflammatory or auto-immune disease
* Suspected or confirmed infectious disease, including HIV, HCV, HBV
* Anti-inflammatory drug treatment or immuno-modulator.
* Multiple pregnancies
* PTL <24 WOA or >34 WOA
* Patient less than 18 years of age.
* Patient not affiliated to social security insurance

Exclusion Criteria for volunteers:

* Pre-existing diabètes
* Morbid obesity (BMI > 35 kg/m2)
* Inflammatory or auto-immune disease
* Suspected or confirmed infectious disease, including HIV, HCV, HBV
* Anti-inflammatory drug treatment or immuno-modulator.
* Minor person
* Person not affiliated to social security insurance
* History of twin pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of women with delivering before 7 days | 7 days
  Main outcome will be a delivery occurring within 7 days post admission for PTL. Women discharged from hospital before day 7 and not having delivered will not be censored; they will be classified as non-delivering before D7.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'investigation clinique plurithématique, Dijon, France

REFERENCES:
- [Result] Bardou M, Hadi T, Mace G, Pesant M, Debermont J, Barrichon M, Wendremaire M, Laurent N, Sagot P, Lirussi F. Systemic increase in human maternal circulating CD14+CD16- MCP-1+ monocytes as a marker of labor. Am J Obstet Gynecol. 2014 Jan;210(1):70.e1-9. doi: 10.1016/j.ajog.2013.08.031. Epub 2013 Aug 29. PMID 23994222
- [Derived] Wendremaire M, Hadi T, Lopez TE, Guy J, Neiers F, Garrido C, Simon E, Jaffal Z, Bernigal V, Bardou M, Lirussi F. Immunophenotyping and Activation Status of Maternal Lymphocytes to Predict Spontaneous Preterm Birth in Women With Threatened Preterm Labor: A Prospective Observational Study. Am J Reprod Immunol. 2024 Dec;92(6):e70015. doi: 10.1111/aji.70015. PMID 39625044